CLINICAL TRIAL: NCT01643902
Title: Safety of Intravenous Thrombolytics in Stroke on Awakening
Acronym: SAIL-ON
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Victor C Urrutia, MD, Associate Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28242
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Stroke
Keywords: Stroke; Wake up; IV tPA; Thrombolytic
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IV tPA (Experimental): Treatment will be initiated within 4.5 hours of awakening, for patients who meet inclusion criteria
  Interventions: Drug: tPA

INTERVENTIONS:
Drug: tPA — IV tPA 0.9 mg/kg maximum of 90 mg. Administered by standard protocol. 10% of the dose by intravenous bolus injection, followed by infusion of the remainder over an hour. Treatment will be initiated within 4.5 hours of awakening with preferred target door to needle time of 60 minutes or less from ED arrival.
  Other Names: Activase; Alteplase

SUMMARY:
The primary objective of this study is to evaluate the safety of intravenous tissue plasminogen activator (IV tPA) in patients waking up with symptoms of acute stroke and presenting to the Emergency Department (ED) within 4.5 hours from awakening, and meeting standard criteria for treatment with IV tPA for acute stroke.

The hypothesis is that patients that wake up with stroke symptoms may have developed the stroke at the time of awakening, and may be within the 4.5 hour window if they arrive to the ED within that time, therefore IV tPA should be safe and effective in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age greater or equal to 18 years, and lower or equal to 80 years.
* Signs and symptoms of acute ischemic stroke.
* Symptoms present upon awakening.
* Arriving to the Emergency Department within 4.5 hours of awakening. Treatment with IV tPA must be initiated prior to 4.5hours from waking up.
* NIHSS >3
* A non-contrast head CT without hemorrhage and without hypodensity more than 1/3 of the middle cerebral artery (MCA) territory; or MRI demonstrating no hemorrhage, and with a diffusion-weighted imaging (DWI) lesion no greater than 70 mL and FLAIR without a well defined hyperintense lesion that is more than 1/3 of the MCA territory.
* Pre-morbid modified Rankin score of 0 or 1.

Exclusion Criteria:

* Rapidly improving deficit to an NIHSS less than 3.
* Sustained systolic blood pressure greater than 185 mmHg or diastolic blood pressure greater than 110 mmHg despite treatment.
* Glucose less than 50 mg/dL.
* Stroke or head trauma within last 3 months.
* History of intracranial hemorrhage. Symptoms of subarachnoid hemorrhage.
* Major surgery within 14 days.
* Gastrointestinal (GI)/Genito-urinary (GU) hemorrhage within 21 days.
* International normalized ratio (INR) > 1.7.
* Heparin within 48 hours with an elevated activated partial thromboplastin time (aPTT).
* Platelet count less than 100,000.
* Presumed septic embolus or suspicion of bacterial endocarditis.
* Suspicion of aortic dissection.
* Use of anticoagulants such as dabigatran, rivaroxaban, apixaban, enoxaparin.
* Pregnant or lactating women.
* Known allergy or sensitivity to tPA.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor C Urrutia, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - The Johns Hopkins Hospital, Baltimore, Maryland

REFERENCES:
- [Derived] Urrutia VC, Faigle R, Zeiler SR, Marsh EB, Bahouth M, Cerdan Trevino M, Dearborn J, Leigh R, Rice S, Lane K, Saheed M, Hill P, Llinas RH. Safety of intravenous alteplase within 4.5 hours for patients awakening with stroke symptoms. PLoS One. 2018 May 22;13(5):e0197714. doi: 10.1371/journal.pone.0197714. eCollection 2018. PMID 29787575

RESULTS

PARTICIPANT FLOW:
Groups:
- IV tPA: Treatment will be initiated within 4.5 hours of awakening, for patients who meet inclusion criteria
  rt-PA: IV rt-PA 0.9 mg/kg minimum of 90 mg. Administered by standard protocol. 10% of the dose by intravenous bolus injection, followed by infusion of the remainder over an hour. Treatment will be initiated within 4.5 hours of awakening with preferred target foor to needle time of 60 minutes or less from ED arrival.
Period: Overall Study
Arm/Group | IV tPA
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- IV tPA: Treatment will be initiated within 4.5 hours of awakening, for patients who meet inclusion criteria
  IV tPA: IV tPA 0.9 mg/kg maximum of 90 mg. Administered by standard protocol. 10% of the dose by intravenous bolus injection, followed by infusion of the remainder over an hour. Treatment will be initiated within 4.5 hours of awakening with preferred target door to needle time of 60 minutes or less from ED arrival.
Arm/Group | IV tPA
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 11
Age, Continuous [Mean (Full Range); unit: years] | 65 [47 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Symptomatic Intracerebral Hemorrhage Within 36 Hours of Treatment
Description: Symptomatic intracerebral hemorrhage by using the European Cooperative Acute Stroke Study (ECASS) 3 criteria as well as the original National Institutes of Neurological Disorders and Stroke (NINDS) Intravenous tissue plasminogen activator (IV tPA) trial criteria for comparison.
  ECASS 3 criteria: hemorrhage in brain imaging, and an increase of 4 or more points on the National Institutes of Health Stroke Scale (NIHSS) from baseline.
  NINDS IV tPA trial criteria: a hemorrhage not seen in previous brain imaging, associated with a neurological decline attributable to the hemorrhage.
Time Frame: within 36 hours of treatment
Population: No symptomatic intracerebral hemorrhage was observed by either NINDS IV tPA trial or ECASS 3 criteria.
Measure: Number; unit: participants
Groups:
- IV Rt-PA: Treatment will be initiated within 4.5 hours of awakening, for patients who meet inclusion criteria
  IV tPA: IV tPA 0.9 mg/kg maximum of 90 mg. Administered by standard protocol. 10% of the dose by intravenous bolus injection, followed by infusion of the remainder over an hour. Treatment will be initiated within 4.5 hours of awakening with preferred target door to needle time of 60 minutes or less from Emergency department (ED) arrival.
Arm/Group | IV Rt-PA
Number analyzed (Participants) | 20
participants | 0

2. Secondary Outcome: Functional Outcome by the Modified Rankin Scale at 90 Days
Description: The modified Rankin scale (mRS) is a scale of disability after stroke, with a range of 0 to 6.
  0, no symptoms at all.
  1. no significant disability despite symptoms; able to carry out all usual duties and activities.
  2. slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance.
  3. moderate disability; requiring some help, but able to walk without assistance.
  4. moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance.
  5. severe disability; bedridden, incontinent and requiring constant nursing care and attention.
  6. dead.
Time Frame: 90 days
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | IV tPA
Number analyzed (Participants) | 20
units on a scale | 1 [0 to 5]

ADVERSE EVENTS:
Arm/Group | IV tPA
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IV tPA (N=20)
Asymptomatic intracerebral hemorrhage (Nervous system disorders) | 2 (2) — Presence of intracranial hemorrhage in routine brain imaging after IV tPA, without any deterioration in neurological status.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No